CLINICAL TRIAL: NCT01957787
Title: Multicenter Study of Metastatic Lung Tumors Targeted by Interventional Cryoablation Evaluation
Brief Title: Study of Cryoablation for Metastatic Lung Tumors
Acronym: SOLSTICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUC13-LNG079
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Neoplasm Metastasis
Keywords: Metastatic lung tumors; Pulmonary metastatic disease
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryoablation (Experimental): Participants will undergo a cryoablation procedure with the Galil Medical Cryoablation System according to the manufacturer's guidelines. Participant preparation, anesthesia, intra-operative monitoring, and postoperative management for the study cryoablation procedure will be identical to those for standard cryoablation treatment routinely performed at the clinical centers that participated in this study and will be at the discretion of the Investigators. Tumors in both lungs are to be treated at an appropriate interval, determined on an individual basis. Treatment of bilateral index tumors in a single treatment session will not be performed. All participants will receive cryoablation of up to 6 metastatic lung tumors. Treatment of all study index tumors are to be completed within an 8-week window.
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Application of extremely cold temperatures to the identified tumor(s).
  Other Names: Cryotherapy; Visual-ICE® Cryoablation System; PresIce® Cryoablation System; SeedNet® Cryoablation System; IceEDGE® 2.4 Cryoablation Needles; IceRod® PLUS Cryoablation Needles; IceSphere™ Cryoablation Needles

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of cryoablation therapy used to treat tumors in participants with pulmonary metastatic disease. This study is to enroll participants who will undergo cryoablation of at least 1 metastatic pulmonary tumor that is less than or equal to 3.5 centimeter (cm). Participants will be followed 24 months post their cryoablation procedure.

DETAILED DESCRIPTION:
Treatment for pulmonary metastatic disease may include surgery, chemotherapy, radiation therapy, or a combination of treatments. However, several variables may exclude participants from these treatments such as multiple tumors, multiple previous surgeries, pulmonary dysfunction, or co-morbid medical conditions. For these participants, percutaneous cryoablation may be a suitable option.

Ablation of metastatic lung tumors is a rapidly expanding area within interventional oncology. Cryotherapy, radiofrequency, laser, and microwave have all been shown to be effective. Cryotherapy offers a wide range of anatomic and tumor treatment options because of the ability to visualize the ice under imaging guidance and the preservation of collagenous tissue structure. Cryoablation has been extensively performed in the prostate and kidney with favorable outcomes reported in the literature. More recently, cryoablation has been shown to be safe in the treatment of lung tumors with CT guidance.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years old.
* Participant has signed a written informed consent.
* Participant presents with Stage 4 pulmonary metastatic disease with metastatic disease previously confirmed by prior biopsy; or Participant presents with Stage 4 pulmonary metastatic disease previously confirmed on imaging (for example, computerized tomography or CT) with histology proven primary cancer.
* Participant has up to 6 local pulmonary metastases targetable by cryoablation.
* Targeted index tumor(s) defined as intra pulmonary or pleural with a maximum size of 3.5 cm, measured in the longest cross-sectional dimension.
* The target index tumor(s) is determined (by CT images) to be in a location where cryoablation is technically achievable based on the proximity of adjacent organs/ structures and is greater than 0.5 cm from any critical organ/structure (possibly achieved with additional maneuvers such as iatrogenic pneumothorax or hydrodissection).
* Karnofsky Performance Scale (KPS) score greater than or equal to 60.
* Platelet count greater than 50,000/millimeters (mm)^3 within 8 weeks prior to initial cryoablation procedure.
* International Normalized Ratio (INR) less than 1.5 within 8 weeks prior to initial cryoablation procedure.
* Participant has a life expectancy of greater than 3 months.

Exclusion Criteria:

* Participant's index tumor(s) is primary lung cancer.
* Participant has uncontrollable primary or metastatic disease outside of the lung.
* Participant is unable to lie flat or has respiratory distress at rest.
* Participant has a coagulopathy or bleeding disorder which is uncontrolled.
* Absolute Neutrophil Count (ANC) <1000 within 8 weeks prior to initial cryoablation procedure.
* Participant has evidence of active systemic, pulmonary, or pericardial infection.
* Participant has a debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment or follow up.
* Participant is currently participating in other experimental studies that could affect the primary endpoint (for example, experimental chemotherapy regimen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry de Baere, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Matthew Callstrom, MD, Study Chair — Mayo Clinic
Locations (10):
- United States (8):
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - Cancer Treatment Centers of America at Southeastern Regional Medical Center, Newnan, Georgia
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Medical Center, New York, New York
  - State University of New York at Stony Brook, Stony Brook, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - Inova Alexandria Hospital CVIR, Alexandria, Virginia
- France (2):
  - Institut Bergonié, Bordeaux, Aquitaine
  - Institut Gustave Roussy, Villejuif, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillams A. Lung tumour ablation - where are we now? Cancer Imaging. 2008 Apr 22;8(1):116-7. doi: 10.1102/1470-7330.2008.0015. PMID 18442957
- [Background] Ahmed A, Littrup P. Percutaneous cryotherapy of the thorax: safety considerations for complex cases. AJR Am J Roentgenol. 2006 Jun;186(6):1703-6. doi: 10.2214/AJR.04.1068. No abstract available. PMID 16714662
- [Background] Kawamura M, Izumi Y, Tsukada N, Asakura K, Sugiura H, Yashiro H, Nakano K, Nakatsuka S, Kuribayashi S, Kobayashi K. Percutaneous cryoablation of small pulmonary malignant tumors under computed tomographic guidance with local anesthesia for nonsurgical candidates. J Thorac Cardiovasc Surg. 2006 May;131(5):1007-13. doi: 10.1016/j.jtcvs.2005.12.051. PMID 16678583
- [Background] Asimakopoulos G, Beeson J, Evans J, Maiwand MO. Cryosurgery for malignant endobronchial tumors: analysis of outcome. Chest. 2005 Jun;127(6):2007-14. doi: 10.1378/chest.127.6.2007. PMID 15947313
- [Background] Wang H, Littrup PJ, Duan Y, Zhang Y, Feng H, Nie Z. Thoracic masses treated with percutaneous cryotherapy: initial experience with more than 200 procedures. Radiology. 2005 Apr;235(1):289-98. doi: 10.1148/radiol.2351030747. PMID 15798173
- [Background] Inoue M, Nakatsuka S, Yashiro H, Ito N, Izumi Y, Yamauchi Y, Hashimoto K, Asakura K, Tsukada N, Kawamura M, Nomori H, Kuribayashi S. Percutaneous cryoablation of lung tumors: feasibility and safety. J Vasc Interv Radiol. 2012 Mar;23(3):295-302; quiz 305. doi: 10.1016/j.jvir.2011.11.019. Epub 2012 Jan 20. PMID 22265246
- [Background] Yamauchi Y, Izumi Y, Kawamura M, Nakatsuka S, Yashiro H, Tsukada N, Inoue M, Asakura K, Nomori H. Percutaneous cryoablation of pulmonary metastases from colorectal cancer. PLoS One. 2011;6(11):e27086. doi: 10.1371/journal.pone.0027086. Epub 2011 Nov 9. PMID 22096520
- [Background] Pusceddu C, Sotgia B, Fele RM, Melis L. CT-guided thin needles percutaneous cryoablation (PCA) in patients with primary and secondary lung tumors: a preliminary experience. Eur J Radiol. 2013 May;82(5):e246-53. doi: 10.1016/j.ejrad.2012.12.010. Epub 2013 Feb 8. PMID 23394762

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Number of Index Tumors
Groups:
- Cryoablation: Participants underwent a cryoablation procedure with the Galil Medical Cryoablation System according to the manufacturer's guidelines. Participant preparation, anesthesia, intra-operative monitoring, and postoperative management for the study cryoablation procedure were identical to those for standard cryoablation treatment routinely performed at the clinical centers that participated in this study and were at the discretion of the Investigators. Tumors in both lungs were to be treated at an appropriate interval, determined on an individual basis. Treatment of bilateral index tumors in a single treatment session was not performed. All participants received cryoablation of up to 6 metastatic lung tumors. Treatment of all study index tumors was completed within an 8-week window.
Period: Overall Study
Arm/Group | Cryoablation
Started | 131; 226 Number of Index Tumors (Participant who was withdrawn prior to study treatment was not included in Number of Index Tumors.)
Intent-to-Treat (ITT) Population (Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed.) | 130; 226 Number of Index Tumors
Modified ITT (mITT) Population (Participants in the ITT population and met all study entry criteria.) | 128; 224 Number of Index Tumors
Completed | 95; 170 Number of Index Tumors
Not Completed | 36; 56 Number of Index Tumors
Not completed — Death | 18
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — Entered Hospice or Similar Program | 2
Not completed — Index Tumor(s) Resected | 2
Not completed — Index Tumor was Primary Lung Cancer | 2
Not completed — Local therapy, not cryoablation | 6

BASELINE CHARACTERISTICS:
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed and met all study entry criteria (mITT population).
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 62
  More than one race | 0
  Unknown or Not Reported | 59
Number of Index Tumors Per Participant [Count of Participants; unit: Participants]
  1 Tumor | 79
  2 Tumors | 23
  3 Tumors | 15
  4 Tumors | 5
  5 Tumors | 2
  6 Tumors | 4

OUTCOME MEASURES:

1. Primary Outcome: Local Tumor Control for Each Index Tumor as Measured by Imaging at Month 12
Description: Local tumor control defined as the absence of local treatment failure 12 months following study cryoablation based on site-reported data. Local control was achieved if the 3-axis measurement (that is, the greatest trans-axial diameter plus the 2 perpendicular diameters) of a tumor at Month 12 was less than 20% larger than the 3-axis measurement of the tumor at Month 1 following study cryoablation. A separate evaluation of local tumor control at Month 12 following cryoablation was completed per index tumor. Month 1 data served as the baseline for this analysis; if Month 1 data was missing, Month 3 data were used. Tumors with a local failure at the prior study visit and those with repeat cryoablation procedures prior to Month 12 were counted as failures. Imaging for assessment of tumor measurements was performed using CT or 18 F-fluorodeoxyglucose positron emission tomography-CT with or without contrast.
Time Frame: Month 1 (Month 3 if Month 1 Data was missing) and Month 12
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed and met all study entry criteria (mITT population). Multiple imputation methods for missing data were applied.
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: Number of Tumors
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
Number analyzed (Number of Tumors) | 224
percentage of tumors | 84.6 [78.6 to 89.2]
Statistical Analysis 1: Comparison: Cryoablation; The null hypothesis was tested comparing the lower bound of the Wald 97.5% 1-sided confidence interval for the estimated rate of local tumor control to the performance goal of 84.0%. If the lower bound was greater than 84.0%, the null hypothesis was rejected and the endpoint was considered met; Test type: Other; p = 0.410, Random effects logistic regression model — Estimates of the log odds and Wald standard error from a random effects logistic regression model were combined across imputed datasets for reference

2. Secondary Outcome: Number of Participants With an Intra- or Post-operative Adverse Event, a Serious Adverse Event, or an Unanticipated Adverse Device Effect
Description: The number of participants with the following categories of adverse events is presented: an intra-operative, a post-operative, a serious adverse event, or an unanticipated adverse device effect. The adverse events that are presented are related to the cryoablation procedure. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to 30 days post-cryoablation
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed (ITT Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 130
Participants
  Intra-operative nonserious adverse event | 39
  Post-operative nonserious adverse event | 18
  Serious adverse events | 15
  Intra-operative serious adverse event | 4
  Post-operative serious adverse event | 4
  Unanticipated adverse device effect | 0

3. Other Pre Specified Outcome: Local Tumor Control for Each Index Tumor at Month 18 and Month 24
Description: Local tumor control defined as the absence of local treatment failure 18 and 24 months following study cryoablation based on site-reported data. Local control was achieved if the 3-axis measurement (that is, the greatest trans-axial diameter plus the 2 perpendicular diameters) of a tumor at Month 12 was less than 20% larger than the 3-axis measurement of the tumor at Month 1 following study cryoablation. A separate evaluation of local tumor control at Month 12 following cryoablation was completed per index tumor. Month 1 data served as the baseline for this analysis; if Month 1 data was missing, Month 3 data were used. Tumors with a local failure at the prior study visit and those with repeat cryoablation procedures prior to Month 12 were counted as failures. Imaging for assessment of tumor measurements was performed using CT or 18 F-fluorodeoxyglucose positron emission tomography-CT with or without contrast.
Time Frame: Month 1 (Month 3 if Month 1 Data was missing), Month 18 and Month 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: Number of Tumors
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
Number analyzed (Number of Tumors) | 224
percentage of tumors
  Month 18 | 82.3 [75.9 to 87.4]
  Month 24 | 75.1 [66.3 to 82.2]

4. Other Pre Specified Outcome: Overall Participant Survival Post-cryoablation
Description: Overall survival rate was defined as the time in days from the first cryoablation procedure to death. Participants who were alive were censored at the date of the last visit.
Time Frame: Up to Month 24
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
percentage of participants
  0-7 Days | 100
  8-30 Days | 100
  31-90 Days | 100
  91-180 Days | 100
  181-365 Days | 97.6
  366-730 Days | 86.6

5. Other Pre Specified Outcome: Time to Metastatic Lung Disease Progression Beyond the Index Tumor(s)
Description: Time to metastatic lung disease progression beyond the index tumor was defined as the time in days from the first cryoablation procedure to metastatic disease beyond the index tumor site. Participants without metastatic lung disease progression were censored at the date of their last visit or their date of death (due to any cause).
Time Frame: Up to Month 24
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
days | 515 [351 to 733]

6. Other Pre Specified Outcome: Time to Overall Cancer Progression
Description: Time to overall cancer progression was defined as the time in days from the first cryoablation procedure to cancer progression (that is, any location of active cancer disease). Participants without cancer progression were censored at the date of their last visit or their date of death (due to any cause).
Time Frame: Up to Month 24
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
days | 173 [103 to 279]

7. Other Pre Specified Outcome: Local Tumor Control With Additional Cryoablation Galil Medical Technology Treatment(s) of a Previously Treated Index Tumor
Description: Local tumor control, defined as absence of local treatment failure 12 months following study cryoablation based on site-reported data, was achieved if 3-axis measurement (that is, greatest trans-axial diameter plus 2 perpendicular diameters) of a tumor at Month 12 was <20% larger than 3-axis measurement of the tumor at Month 1 following study cryoablation. Separate evaluation of local tumor control at Month 12 following cryoablation was completed per index tumor. Follow-up visits were re-started after additional treatment, per study protocol and continued through the Month 24 visit after the last study cryoablation. Month 1 data served as baseline for analysis; if Month 1 data was missing, Month 3 data were used. Tumors with a local failure at prior study visit and with repeat cryoablation procedures prior to Month 12 were counted as failures. Tumor measurement imaging performed using CT or 18 F-fluorodeoxyglucose positron emission tomography-CT with or without contrast.
Time Frame: Up to Month 12
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed and met all study entry criteria (mITT population) and underwent an additional Cryoablation Galil Medical Technology Treatment.
Measure: Number; unit: percentage of tumors
Units Other Than Participants: Number of Tumors
Arm/Group | Cryoablation
Number analyzed (Participants) | 13
Number analyzed (Number of Tumors) | 16
percentage of tumors | 100

8. Other Pre Specified Outcome: Time to Untreatable Metastatic Lung Disease Control With Cryoablation (Free From Metastatic Lung Disease)
Description: Time to untreatable metastatic lung disease control with cryoablation is defined as the time in days from the first cryoablation procedure to the time when the metastatic lung disease cannot be treated with cryoablation. The percentage of participants free from metastatic disease that is untreatable with cryoablation at the intervals of time of Days 181 to 365 and Days 495 to 730 is presented.
Time Frame: Month 12 (Days 181-365) and Month 24 (Days 495-730)
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed and met all study entry criteria (mITT population) with available data at the respective time point.
Measure: Number; unit: percentage of participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
percentage of participants
  Month 12 (Days 181-365): number analyzed (Participants) | 111
  Month 12 (Days 181-365) | 83.3
  Month 24 (Days 495-730): number analyzed (Participants) | 84
  Month 24 (Days 495-730) | 72.2

9. Other Pre Specified Outcome: Time to Untreatable Metastatic Lung Disease Control With Focal Therapy (Free From Metastatic Lung Disease)
Description: Time to untreatable metastatic lung disease control with focal therapy defined as the time in days from the first cryoablation procedure to the time when the metastatic lung disease cannot be treated by focal (for example, ablation, surgery, SBRT) intervention for control of metastatic lung disease. The percentage of participants free from metastatic disease that is untreatable with focal therapy at the intervals of time of Days 181 to 365 and Days 495 to 730 is presented.
Time Frame: Month 12 (Days 181-365) and Month 24 (Days 495-730)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
percentage of participants
  Month 12 (Days 181-365): number analyzed (Participants) | 109
  Month 12 (Days 181-365) | 81.7
  Month 24 (Days 495-730): number analyzed (Participants) | 83
  Month 24 (Days 495-730) | 72.4

10. Other Pre Specified Outcome: Cryoablation Technical Success at Month 1
Description: A technically successful treatment was defined by the presence of an ablation zone, ground glass opacity, or frank consolidation encompassing the targeted index tumor(s) at no later than the 1 month follow up visit after the cryoablation procedure. Technical success rates and 95% confidence intervals (CIs) were calculated using random effects logistic regression on a tumor level.
Time Frame: Up to Month 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: Number of Tumors
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
Number analyzed (Number of Tumors) | 224
percentage of tumors | 97.2 [93.3 to 98.9]

11. Other Pre Specified Outcome: Change From Baseline in Physical Function as Assessed by the Karnofsky Performance Status (KPS) Scale at Months 1, 3, 6, 12, 18, and 24
Description: The KPS scale is a standard way of measuring the ability of cancer participants to perform ordinary tasks. KPS may be used to determine a participant's prognosis and to measure changes in a participant's ability to function. Assessments were made by examining the change in the baseline scores to those reported post-operatively. KPS scores range from 0 to 100. A higher score means the participant is better able to carry out daily activities.
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 12, Month 18, and Month 24
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed and met all study entry criteria (mITT population) and evaluable KPS scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
units on a scale
  Month 1: number analyzed (Participants) | 123
  Month 1 | -1.14 (6.80)
  Month 3: number analyzed (Participants) | 119
  Month 3 | -1.34 (8.12)
  Month 6: number analyzed (Participants) | 111
  Month 6 | -1.08 (8.35)
  Month 12: number analyzed (Participants) | 102
  Month 12 | -1.86 (8.64)
  Month 18: number analyzed (Participants) | 89
  Month 18 | -3.82 (12.29)
  Month 24: number analyzed (Participants) | 78
  Month 24 | -5.00 (16.02)

12. Other Pre Specified Outcome: Change From Baseline in Quality of Life Over Time as Assessed by the Short Form-12 (SF-12) Generic Measure at Month 1 and Month 3
Description: The SF-12 is a shortened version of the well-known SF-36. The SF-12 assesses 8 domains (physical functioning, role limitations due to physical health problems, bodily pain, social functioning, general mental health, role limitations due to emotional problems, vitality, general health perception). The shorter instrument provides a general measurement of quality of life. Assessments were made by examining the change in the baseline scores to those reported post-operatively. The scores range from 0 to 100. A higher value indicates a better quality of life of the participant.
Time Frame: Baseline, Month 1 and Month 3
Population: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed and met all study entry criteria (mITT population) and evaluable SF-12 scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 128
units on a scale
  Physical Functioning, Month 1: number analyzed (Participants) | 123
  Physical Functioning, Month 1 | -3.9 (28.5)
  Physical Functioning, Month 3: number analyzed (Participants) | 116
  Physical Functioning, Month 3 | -3.2 (28.7)
  Role Physical, Month 1: number analyzed (Participants) | 123
  Role Physical, Month 1 | 1.6 (34.3)
  Role Physical, Month 3: number analyzed (Participants) | 115
  Role Physical, Month 3 | 3.9 (35.9)
  Bodily Pain, Month 1: number analyzed (Participants) | 122
  Bodily Pain, Month 1 | -1.6 (26.6)
  Bodily Pain, Month 3: number analyzed (Participants) | 114
  Bodily Pain, Month 3 | -2.4 (26.4)
  Social Functioning, Month 1: number analyzed (Participants) | 123
  Social Functioning, Month 1 | 3.3 (23.7)
  Social Functioning, Month 3: number analyzed (Participants) | 116
  Social Functioning, Month 3 | 0.9 (29.1)
  Mental Health, Month 1: number analyzed (Participants) | 123
  Mental Health, Month 1 | 2.9 (20.1)
  Mental Health, Month 3: number analyzed (Participants) | 116
  Mental Health, Month 3 | 3.0 (23.1)
  Role Emotional, Month 1: number analyzed (Participants) | 123
  Role Emotional, Month 1 | -2.0 (25.8)
  Role Emotional, Month 3: number analyzed (Participants) | 115
  Role Emotional, Month 3 | 2.6 (24.8)
  Vitality, Month 1: number analyzed (Participants) | 122
  Vitality, Month 1 | -2.7 (29.4)
  Vitality, Month 3: number analyzed (Participants) | 113
  Vitality, Month 3 | -1.3 (29.7)
  General Health Perception, Month 1: number analyzed (Participants) | 123
  General Health Perception, Month 1 | -2.3 (25.1)
  General Health Perception, Month 3: number analyzed (Participants) | 116
  General Health Perception, Month 3 | -2.2 (23.7)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 24
Description: Participants for whom cryoablation via Galil Medical Cryoablation System was attempted or performed (ITT Population).
Arm/Group | Cryoablation
All-Cause Mortality (participants affected / at risk) | 18/130
Serious Adverse Events (participants affected / at risk) | 18/130
Other Adverse Events (participants affected / at risk) | 70/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoablation (N=130)
Coronary artery disease (Cardiac disorders) | 1
Gait imbalance (General disorders) | 1
Abdominal infection (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9
Gaseous embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoablation (N=130)
Sinus tachycardia (Cardiac disorders) | 1
Abdominal distention (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bilateral leg edema (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain at needle site (General disorders) | 12
Allergic reaction (Immune system disorders) | 1
Device related infection (Infections and infestations) | 1
Hepatic infection (Infections and infestations) | 1
MRSA infected decubitus ulcer (Infections and infestations) | 1 — Methicillin-resistant Staphylococcus aureus (MRSA)
Oropharyngeal candidiasis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Burn (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Steroid induced hyperglycemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Paresthesia (Nervous system disorders) | 1
Radiculitis (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Diaphragm paralysis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Left-sided pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 39
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash on face and abdomen (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Galil Medical can require Investigator to postpone publications/presentations for up to 12 months so data from all sites can be published. Galil Medical will limit review of Investigator's draft to confirm Confidential Information is not being disclosed. If Galil Medical notes publishing Study results may affect obtaining a patent, Investigator may not publish for up to 60 days until patent application is filed. Investigator will acknowledge Galil Medical in any publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2014-02-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT01957787/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT01957787/SAP_001.pdf